CLINICAL TRIAL: NCT05825105
Title: Efectividad Del Plasma Rico en Plaquetas (PRP) Para la disminución Objetiva Del Dolor y la recuperación Funcional Del Miembro Inferior en Osteoartritis de Rodilla. Evaluación de Alternativas metodológicas
Brief Title: Effectiveness of Platelet-rich Plasma Treatment of Knee Osteoarthritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad Nacional de Entre Rios (Other)
Collaborators: National Council of Scientific and Technical Research, Argentina (Other Government)
Responsible Party: Principal Investigator, Pablo Schierloh, Associate Investigator, Universidad Nacional de Entre Rios
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRP-BXD1; IS004027 (Other: RENIS)
Record Dates: First submitted 2023-03-28; First posted 2023-04-24 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Knee Osteoarthritis
Keywords: Autologous Treatments; Public Health; Lower Extremity; Argentina; Real-world studies
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP-1 (Experimental): Platelet-rich plasma, short treatment (three sessions every two weeks)
  Interventions: Biological: Platelet-Rich Plasma
- PRP-2 (Active Comparator): Platelet-rich plasma, long treatment (three sessions every four weeks)
  Interventions: Biological: Platelet-Rich Plasma

INTERVENTIONS:
Biological: Platelet-Rich Plasma — The PRP will be prepared using a single centrifugation process. Approximately 30 ml of peripheral blood will be drawn and collected into a vacutainer tubes with sodium citrate anticoagulant 0.129 mol/l (3.8%). The tubes will then be centrifuged at 900 RPM for 12 minutes at room temperature in a benchtop centrifuge. We will separate the lower third of the plasma fraction from all tubes with a syringe and needle, taking care to avoid the leukocyte layer. The PRP will be refrigerated at 4°C for no less than 1 hour. We will not use any exogenous factors to stimulate the platelet activation process. The periauricular skin surface will be disinfected with a povidone iodine solution, and an intra-articular local anesthetic with 1% lidocaine will be applied. A 21-gauge needle will be placed at the point of application. Finally, PRP will be injected into the joint, and the needle will be removed.

SUMMARY:
Osteoarthritis (OA) is a disease that affects the joints of the body, causing pain, stiffness, and reduced mobility. To treat knee OA, a therapy called platelet-rich plasma (PRP) is used, which involves making a concentrated substance from the patient's own blood and injecting it into the joint. It has been shown that this therapy is effective in reducing pain; however, more research is needed to optimize the preparation and identify which patients are more receptive to the treatment. The primary objective of this study is to evaluate two modalities of PRP application and determine whether these treatments result in better pain reduction and improved functionality. The secondary objective is to explore the association between changes in LEFS questionnaire scores and/or maximal quadriceps isometric strength and possible clinical improvement.

ELIGIBILITY:
Inclusion Criteria:

* Radiological diagnosis of knee OA
* Age over 35 years old
* WOMAC value of 24 or higher at the time of recruitment

Exclusion Criteria:

* Patients with knee prosthesis, rheumatoid arthritis, contralateral lower limb amputation, any type of blood dyscrasia, hypofibrinogenemia, depot pool syndrome, or any other form of thrombocytopathy or chronic leukocytosis will be excluded from the study.
* Patients with anticoagulant or acute coagulopathies, as well as carriers of any infectious disease or superficial infection at the puncture site, will be temporarily excluded from the study until their clinical recovery is confirmed by laboratory testing.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change in the Western Ontario and McMaster Universities (WOMAC) Ostearthritis Index | Baseline, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 24 weeks, 48 weeks.
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) questionnaire assesses the symptoms and physical disability of individuals with OA. The WOMAC consists of multiple-choice questions, and the responses are scored from zero to four. The final score is calculated between 0 and 96, where higher scores correspond to greater pain, stiffness, and lower functionality, indicating worsening symptoms.

SECONDARY OUTCOMES:
Change in the the Lower Extremity Functional Scale (LEFS) Index | Baseline, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 24 weeks, 48 weeks.
  The Lower Extremity Functional Scale (LEFS) questionnaire is a self-administered questionnaire assessing functional status in patients with various lower limb musculoskeletal conditions, including OA. It consists of 20 items, each scored on a 5-point scale. The maximum possible score is 80, indicating the best functional level.
Change in Maximum Voluntary Isometric Contraction (MVIC) strength of the quadriceps | Baseline, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 24 weeks, 48 weeks.
  MVIC (maximum voluntary isometric contraction) strength of the quadriceps will be assessed using an instrumented load cell, which measures in kilograms. Objective and reliable assessment of muscle strength is well-supported for monitoring disease progression and evaluating therapeutic interventions. The test will involve asking the patient to extend the knee with maximum possible force for 3 seconds, ensuring that the hip and knee are at 90 degrees. Three repetitions will be performed with 2-minute rests.
Centre of pressure (COP) on the plantar surface of the foot | Baseline, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 24 weeks, 48 weeks.
  The measurement of plantar pressure pattern and COP will be performed using a foot-X AR-1 pressure platform. The patient will be positioned upright or anatomically on the platform for a period of time during which the application will record the pressure values. The measurement will be bipedal (both feet on the platform), so both an integral COP of both feet and an individual COP of each foot will be obtained.
Timed Up and Go (TUG) Test | Baseline, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 24 weeks, 48 weeks.
  The FTSTS and TUG tests are reliable and validated clinical tools that are used as predictors of health problems or disability. The first one consists of the time it takes to sit and stand five times in a row. The second one is similar, but adds a walk at a certain distance.
Five Times Sit to Stand (FTSTS) Test | Baseline, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 24 weeks, 48 weeks.
  The FTSTS and TUG tests are reliable and validated clinical tools that are used as predictors of health problems or disability. The first one consists of the time it takes to sit and stand five times in a row. The second one is similar, but adds a walk at a certain distance.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Research and Development in Bioengineering and Bioinformatics (IBB-CONICET-UNER), Oro Verde, Entre Ríos Province, Argentina

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
URL: https://osf.io/nkm3v/?view_only=4e754432fbd644948b07c39554d7dba6